CLINICAL TRIAL: NCT06941935
Title: Etiological Classification-guided Individual Intervention in Primary Hypertension: An All-comer Registry Study
Brief Title: Etiological Classification-guided Individual Intervention in Primary Hypertension
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, professor of Medicine, Shanghai 10th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GENESIS
Record Dates: First submitted 2025-04-13; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Hypertension
Keywords: Etiological Classification; Digital Intervention
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hypertension precision diagnosis and treatment group (Experimental): participants will undergo etiological testing for primary hypertension, followed by tailored pharmacological treatment and digital blood pressure monitoring, with regular medication adjustments.
  Interventions: Other: Etiological Classification and Digital Intervention

INTERVENTIONS:
Other: Etiological Classification and Digital Intervention — Eligible participants will first undergo a 1-week home blood pressure diary and 24-hour ambulatory blood pressure assessment. After a confirmed diagnosis of hypertension, etiological subtyping will be performed. Based on the blood pressure evaluation results and etiological classification, the most appropriate antihypertensive medication will be selected. Simultaneously, a personalized lifestyle prescription will be provided according to the patient's individual circumstances. Following medication initiation, participants will continue to monitor their blood pressure through home diaries. Monthly evaluations will be conducted, and if blood pressure fails to reach the target value, medication adjustments will be made based on the blood pressure diary until target levels are achieved. This regimen will be maintained long-term.

SUMMARY:
Eligible participants will first undergo a 1-week home blood pressure diary and 24-hour ambulatory blood pressure assessment. After a confirmed diagnosis of hypertension, etiological subtyping will be performed. Based on the blood pressure evaluation results and etiological classification, the most appropriate antihypertensive medication will be selected. Simultaneously, a personalized lifestyle prescription will be provided according to the patient's individual circumstances. Following medication initiation, participants will continue to monitor their blood pressure through home diaries. Monthly evaluations will be conducted, and if blood pressure fails to reach the target value, medication adjustments will be made based on the blood pressure diary until target levels are achieved. This regimen will be maintained long-term.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years.
* Diagnosed primary hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg).
* signed informed consent.

Exclusion Criteria:

* Secondary hypertension or arrhythmias affecting blood pressure accuracy (e.g., atrial fibrillation).
* Comorbidities such as diabetes, chronic kidney disease (eGFR < 30 mL/min/1.73m²), coronary artery disease, heart failure, or serious valvular heart disease.
* History of stroke or myocardial infarction.
* Pregnancy, breastfeeding, or planning to become pregnant.
* Life expectancy < 1 year.
* Participation in another clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Blood Pressure Recorded in a 1-Week Home Blood Pressure Diary | 3 months following intervention
  Changes in blood pressure recorded (SBP/DBP) in a 1-week home blood pressure diary from baseline to 3 months.

SECONDARY OUTCOMES:
Change in 24-hour Ambulatory Blood Pressure Monitoring | 1/2/3 months following intervention
  Change in 24-hour ambulatory blood pressure monitoring (daytime, nighttime, and overall SBP/DBP) at 1/2 /3 months.
Change in Home Blood Pressure Monitoring | 1/2 months following intervention
  Change in home blood pressure monitoring (SBP/DBP) at 1/2months.
Control Rate | 3 months following intervention
  Proportion of patients achieving target blood pressure at 3 months.
Drug adjustment times | 3 months following intervention
  The total number of times to adjust blood pressure medication in 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Cardiology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality